CLINICAL TRIAL: NCT02356705
Title: Intranasal Midazolam in Children as a Pre-Operative Sedative - Part 2
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Jennifer Victory, RN, CCRC (Other)
Responsible Party: Sponsor-Investigator, Jennifer Victory, RN, CCRC, Clinical Research Nurse Supervisor, Bassett Healthcare
Organization: Bassett Healthcare (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1098
Record Dates: First submitted 2015-02-02; First posted 2015-02-05 (Estimated); Results first posted 2021-02-25 (Actual); Last update posted 2022-03-16 (Actual); Status verified 2022-03

CONDITIONS: Sedation
MeSH Terms: interventions — Midazolam; Lidocaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Saline Placebo (Placebo Comparator): Control patients will receive intranasal saline
  Interventions: Drug: saline placebo
- Nasal Midazolam Only (Active Comparator): Patients will receive 0.2 mg/kg of intranasal midazolam
  Interventions: Drug: Midazolam
- Midazolam Plus Xylocaine (Active Comparator): Patients will receive 0.2 mg/kg intranasal midazolam plus xylocaine 4% in a dose based on 50% of the volume of the midazolam.
  Interventions: Drug: Midazolam; Drug: xylocaine

INTERVENTIONS:
Drug: Midazolam — midazolam 0.2 mg/kg given intranasally
  Arms: Midazolam Plus Xylocaine; Nasal Midazolam Only
Drug: xylocaine — intransal xylocaine given in conjunction with intranasal midazolam
  Arms: Midazolam Plus Xylocaine
Drug: saline placebo — intranasal saline given as placebo
  Arms: Saline Placebo

SUMMARY:
Midazolam is often given before surgery to sedate a patient before anesthesia is given. Children are often given a small dose either by mouth or squirted into the nose. Children will often spit out the oral midazolam, making it difficult to know how much medicine, if any, they have received. Giving midazolam into the nose is more reliable, but children may complain of pain, stinging, and may become upset due to the discomfort. Nosebleeds may also occur when midazolam is squirted alone into the nose. The purpose of this study is to see if adding a numbing medicine, xylocaine, to the nasal midazolam makes giving the midazolam easier and more comfortable without affecting how the midazolam works as a sedative. This is follow up to the pilot study, Project # 994. This will expand the previous study, with additional participants and revised xylocaine concentration

ELIGIBILITY:
Inclusion Criteria:

1. Children aged 18 months-7 years, scheduled for a minor Ear/Nose/Throat surgical procedure requiring mask anesthesia
2. American Society of Anesthesiologists (ASA) Class 1 or 2
3. Parent willing and able to provide written informed consent
4. Parent willing and able to complete the Observed Behavioral Distress (OBD) Visual Assessment Scale (VAS)

Exclusion Criteria:

1. ASA Class 3 or greater
2. History of allergy to midazolam or xylocaine
3. Presence of acute respiratory infection at time of surgery
4. Parent unwilling or unable to provide informed consent
5. Parent unwilling or unable to complete the OBD VAS

Ages: 18 Months to 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 42 (Actual)
Dates: Start 2015-01; Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: david Ullman, MD, Principal Investigator — Bassett Healthcare
Locations (1):
- Bassett Healthcare Network, Cooperstown, New York, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Saline Placebo | Nasal Midazolam Only | Midazolam Plus Xylocaine
Started | 14 | 14 | 14
Completed | 14 | 14 | 14
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Saline Placebo | Nasal Midazolam Only | Midazolam Plus Xylocaine | Total
Number analyzed (Participants) | 14 | 14 | 14 | 42
Age, Continuous [Mean (Standard Deviation); unit: years] | 2.4 (1.7) | 3.1 (1.5) | 2.5 (1.7) | 2.7 (1.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 5 | 10 | 22
  Male | 7 | 9 | 4 | 20
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 14 | 14 | 14 | 42

OUTCOME MEASURES:

1. Primary Outcome: Pediatric Pre-Induction Anesthesia Scale at Time of Mask Placement
Description: Pediatric Response to Mask Placement Scale - scaled scored by the anesthesiologist or certified nurse anesthetist (CRNA) at the time of mask placement
  * 1. Agitated: Previous criteria and/or refuses mask. (worst score)
  * 2. Alert: Previous criteria and/or initially refuses mask, but accept after persuasion.
  * 3. Calm: Previous criteria and accepts mask.
  * 4. Drowsy: Previous criteria and accepts mask.
  * 5. Asleep: Previous criteria and accepts mask. (best score)
Time Frame: 25 minutes
Measure: Count of Participants; unit: Participants
Arm/Group | Saline Placebo | Nasal Midazolam Only | Midazolam Plus Xylocaine
Number analyzed (Participants) | 14 | 14 | 14
Participants
  Agitated | 11 | 3 | 6
  Alert | 1 | 1 | 3
  Calm | 2 | 10 | 4
  Drowsy | 0 | 0 | 1
  Asleep | 0 | 0 | 0
Statistical Analysis 1: Comparison: Saline Placebo vs Nasal Midazolam Only vs Midazolam Plus Xylocaine; Test type: Superiority; p = 0.39, Chi-squared

2. Secondary Outcome: Pediatric Pre-Induction Anesthesia Scale at Arrival to Operating Room
Description: Pediatric Pre-Induction Anesthesia Scale - scored by the anesthesiologist or the CRNA upon arrival to the operating room, prior to induction of anesthesia
  * 1. Agitated: Patient clinging to parents and/or crying (worst score)
  * 2. Alert: Patient is aware but not clinging to parent, may whimper but not cry.
  * 3. Calm: Sitting or lying comfortably with spontaneous eye opening.
  * 4. Drowsy: Sitting or lying comfortably with eyes closed, but responding to minor stimulation.
  * 5. Asleep: Eyes closed, arousable but does not respond to minor stimulation. (best score)
Time Frame: 20 minutes
Measure: Count of Participants; unit: Participants
Arm/Group | Saline Placebo | Nasal Midazolam Only | Midazolam Plus Xylocaine
Number analyzed (Participants) | 14 | 14 | 14
Participants
  Agitated | 5 | 1 | 1
  Alert | 1 | 3 | 3
  Calm | 8 | 9 | 9
  Drowsy | 0 | 1 | 1
  Asleep | 0 | 0 | 0
Statistical Analysis 1: Comparison: Saline Placebo vs Nasal Midazolam Only vs Midazolam Plus Xylocaine; Test type: Superiority; p = 0.39, Chi-squared

3. Other Pre Specified Outcome: Time to Discharge
Description: The time (in minutes) from release from the operating room to discharge home
Time Frame: approximately 3 hours
Measure: Median (Inter-Quartile Range); unit: minutes
Arm/Group | Saline Placebo | Nasal Midazolam Only | Midazolam Plus Xylocaine
Number analyzed (Participants) | 14 | 14 | 14
minutes | 35 [29 to 44] | 39.5 [22 to 50] | 35.5 [31 to 45]
Statistical Analysis 1: Comparison: Saline Placebo vs Nasal Midazolam Only vs Midazolam Plus Xylocaine; Test type: Superiority; p = 0.88, Kruskal-Wallis

4. Other Pre Specified Outcome: Number of Participants With Nosebleeds From Time of Drug Administration to Discharge Home
Description: Number of participants with nosebleeds recorded in the pre-operative, intra-operative and post-operative record after study drug administration.
Time Frame: approximately 3 hours
Measure: Count of Participants; unit: Participants
Arm/Group | Saline Placebo | Nasal Midazolam Only | Midazolam Plus Xylocaine
Number analyzed (Participants) | 14 | 14 | 14
Participants | 0 | 0 | 0

5. Other Pre Specified Outcome: Observational Distress Score at 1 Minute (Blinded Study Nurse Assessment)
Description: Visual analog scale measured from 0cm (no distress) to 10cm (high level of distress). Recorded by the blinded study nurse.
Time Frame: 1 minute
Measure: Median (Inter-Quartile Range); unit: cm VAS
Arm/Group | Saline Placebo | Nasal Midazolam Only | Midazolam Plus Xylocaine
Number analyzed (Participants) | 14 | 14 | 14
cm VAS | 0.02 [0 to 0.1] | 0.3 [0.1 to 0.6] | 0.4 [0.01 to 0.6]
Statistical Analysis 1: Comparison: Saline Placebo vs Nasal Midazolam Only vs Midazolam Plus Xylocaine; Test type: Superiority; p = 0.01, Kruskal-Wallis

6. Other Pre Specified Outcome: Observational Distress Score 5 Min (Blinded Study Nurse Assessmnet)
Description: Visual analog scale measured from 0cm (no distress) to 10cm (high level of distress) as measured by the blinded study nurse.
Time Frame: 5minutes
Measure: Median (Inter-Quartile Range); unit: cm VAS
Arm/Group | Saline Placebo | Nasal Midazolam Only | Midazolam Plus Xylocaine
Number analyzed (Participants) | 14 | 14 | 14
cm VAS | 0 [0 to 0.02] | 0.02 [0 to 0.2] | 0 [0 to 0.01]
Statistical Analysis 1: Comparison: Saline Placebo vs Nasal Midazolam Only vs Midazolam Plus Xylocaine; Test type: Superiority; p = 0.08, Kruskal-Wallis

ADVERSE EVENTS:
Time Frame: During patient recovery - from time of entry into the recovery room until discharge (~3 hours)
Arm/Group | Saline Placebo | Nasal Midazolam Only | Midazolam Plus Xylocaine
All-Cause Mortality (participants affected / at risk) | 0/14 | 0/14 | 0/14
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/14 | 0/14
Other Adverse Events (participants affected / at risk) | 0/14 | 0/14 | 0/14

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol (2014-12-05): https://cdn.clinicaltrials.gov/large-docs/05/NCT02356705/Prot_000.pdf